CLINICAL TRIAL: NCT01527669
Title: The Pharmacokinetic Study of Red Yeast Rice Capsule Compared to Lovastatin Tablet in Healthy Subjects.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 201110011MB
Record Dates: First submitted 2012-01-12; First posted 2012-02-07 (Estimated); Last update posted 2012-07-11 (Estimated); Status verified 2012-02

CONDITIONS: Healthy Subjects
Keywords: Red yeast rice; lovastatin; Pharmacokinetics
MeSH Terms: interventions — Lovastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- LipoCol Forte capsules (Experimental): The pharmacokinetic study of red yeast rice capsule compared to lovastatin tablet in healthy subjects.
  Interventions: Drug: LipoCol Forte capsules
- Lovastatin Tablet (Experimental): The pharmacokinetic study of red yeast rice capsule compared to lovastatin tablet in healthy subjects.
  Interventions: Drug: Lovastatin Tablet

INTERVENTIONS:
Drug: LipoCol Forte capsules — The pharmacokinetic study of red yeast rice capsule compared to lovastatin tablet in healthy subjects.
  Arms: LipoCol Forte capsules
Drug: Lovastatin Tablet — The pharmacokinetic study of red yeast rice capsule compared to lovastatin tablet in healthy subjects.
  Arms: Lovastatin Tablet

SUMMARY:
The objective of the study is to evaluate the pharmacokinetics of lovastatin and lovastatin acid of four 600 mg LipoCol Forte capsules compared to that of one 20 mg lovastatin Tablet after single oral administration in healthy subjects.

DETAILED DESCRIPTION:
This study is two-ways crossover design. The subjects will receive a dose of four 600 mg LipoCol Forte Capsules or 20 mg Mevacor Tablet in fasted state in the morning. There is a minimum of a 6-days washout period before crossover of treatments.

Each subject will be admitted before administration of the investigational product in each period. Study responsible personnel will give the subjects a single tablet or four capsules in fasted state in the morning. The blood samples will be drawn prior to the dosing, and 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8 and 12 hours after the dosing.

Observations will be conducted up to 12 hours after the dosing. If no particular health abnormalities are observed in each period, the subjects will be discharged on 12 hours after the dosing.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must be at the age of 20-40 years old and be able to sign informed consent prior to study.
2. Body weight must be above 45 kilograms (kg) and within -20 to +20% of ideal body weight.
3. No clinically significant abnormalities were judged by the principal investigator based on the medical history, physical examination, electrocardiogram, chest X-ray, and routine laboratory evaluations.

Exclusion Criteria:

1. Use of any prescription medication, over-the-counter medications or vitamins within 14 days prior to dosing.
2. Participation in any clinical investigation within 2 months prior to dosing or longer as required by local regulation.
3. Donation or loss of more than 500 milliliter (mL) blood within 3 months prior to dosing.
4. Presence of liver disease (Glutamic Oxaloacetic Transaminase (GOT), Glutamic Pyruvic Transaminase (GPT) or Total-bilirubin greater than 2-fold normal values) or renal disease (blood urea nitrogen (BUN) or creatinine greater than 1.5-fold normal values).
5. Creatine kinase (CK) value greater than 1.5-fold normal value.
6. A known hypersensitivity to statins or their analogs.
7. Permanent confinement to an institution.
8. Individuals are judged by the investigator or co-investigator to be undesirable as subjects for other reasons.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2012-02; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Evaluation of the pharmacokinetic parameters of lovastatin and lovastatin acid in healthy subjects | 1 weeks
  Plasma concentrations of lovastatin and lovastatin acid were detected at following time: (Pre-dose (T0), and 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, and 12 hours after oral administration red yeast rice capsule (LipoCol Forte)or lovastatin. All pharmacokinetic parameters were determined with lovastatin and lovastatin acid concentrations by non-compartment methods.

SECONDARY OUTCOMES:
The incidence rate of adverse event | 1 weeks
  The incidence rate of adverse event

CONTACTS AND LOCATIONS:
Overall Officials: Jyh-Chin Yang, M.D. Ph.D, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

REFERENCES:
- [Derived] Chen CH, Yang JC, Uang YS, Lin CJ. Improved dissolution rate and oral bioavailability of lovastatin in red yeast rice products. Int J Pharm. 2013 Feb 28;444(1-2):18-24. doi: 10.1016/j.ijpharm.2013.01.028. Epub 2013 Jan 23. PMID 23352857